CLINICAL TRIAL: NCT06172361
Title: Efficacy and Safety of Induction and Tapering Therapy With Tofacitinib and Glucocorticoid in Patients With Polymyalgia Rheumatica (ITTG PMR): An Open-label 52-week Randomized Controlled Trial
Brief Title: Induction and Tapering Therapy With Tofacitinib and Glucocorticoid in Patients With Polymyalgia Rheumatica
Acronym: ITTGPMR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weiqian Chen, Clinical Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20230087C-X1
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica; Tofacitinib; Glucocorticoid
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Prednisone; prednylidene

STUDY DESIGN:
Intervention Model Description: Treatment group: Prednisone (or equivalent dose of methylprednisolone) + Tofacitinib
  Positive control group: prednisone (or equivalent dose of methylprednisolone)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Prednisone (or equivalent dose of methylprednisolone) + Tofacitinib
  Interventions: Drug: Prednisone+Tofacitinib
- Positive control group (Active Comparator): prednisone (or equivalent dose of methylprednisolone)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone+Tofacitinib — Withdrawal of prednisone (or equivalent dose of methylprednisolone) within 4 weeks: 5mg tid for 2 weeks, 5mg bid for 1 week, 5mg qd for 1 week, then discontinue.
  Take Tofacitinib 10mg/d for 3 months, then 7.5mg/d for 2 months, followed by 5mg qd for 2 months, then 5mg qod for 2 months, and finally 5mg every 3 days for 2 months, discontinue the Tofacitinib for 1 month. If there is a relapse during the dose reduction process, resume Tofacitinib at the original dosage.
  Other Names: Pred+Tof
  Arms: Treatment group
Drug: Prednisone — Prednisone 15mg (or equivalent dose of methylprednisolone) was set as the initial treatment of PMR. When improvement was achieved, the dose of Prednisone was reduced to 10mg daily within 4-10 weeks; When remission was achieved, then taper Prednisone gradually by 2.5mg every 6-8 weeks. Once relapse occurred, the dose increased to the pre-relapse dose. If reducing pred dosage is difficult, Methotrexate (MTX) 10mg qw can be added after 24 weeks.
  Other Names: Pred
  Arms: Positive control group

SUMMARY:
This will be efficacy and safety of Induction and Tapering Therapy with Tofacitinib and Glucocorticoid in patients with Polymyalgia Rheumatica (ITTG PMR): An open-label 52-week randomized controlled trial

DETAILED DESCRIPTION:
Rheumatic polymyalgia (PMR) is more commonly observed in individuals over the age of 50, who may have a higher prevalence of osteoporosis, diabetes, cardiovascular diseases, and other chronic conditions. Currently, glucocorticoids are the primary treatment for PMR, but they can lead to various side effects, and recurrence is common during steroid tapering. Our previous 24-week study confirmed the effective treatment of PMR patients with tofacitinib. Given the relatively slow efficacy of tofacitinib, early adjunctive therapy with NSAIDs is needed. To address this, we are planning an open-label 52-week randomized controlled trial. This study aims to assess the use of tofacitinib in combination with glucocorticoids to induce rapid improvement, followed by rapid tapering of steroids and slow tapering of tofacitinib. The objective is to observe the efficacy and safety of this regimen for PMR, providing a new treatment option for clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. PMR patients who fulfilled the 1982 Chuang criteria or 2012ACR/EULAR criteria for PMR; They did not receive any glucocorticoids or biological agents during the 2 weeks period that preceded their inclusion in the study;
2. Patients with high activity rheumatic polymyalgia: disease activity score PMR-AS (Table 3) > 10,
3. Adults age 50-88, Weight 45-85Kg,
4. ESR>20mm/h or CRP >50mg/L (5mg/dl),
5. Informed consent.

Exclusion Criteria:

1. Patients with known allergies to tofacitinib, prednisone or methylprednisolone,
2. Patients with identified giant cell arteritis, systemic lupus erythematosus, rheumatoid arthritis, calcium pyrophosphate deposition (CPPD) arthropathy, and other rheumatic diseases,
3. Patients with severe osteoarthritis,
4. Subjects with any severe acute, chronic or recurrent infection (e.g. pneumonia or pyelonephritis, recurrent pneumonia, chronic bronchiectasis, tuberculosis, etc.),
5. Hepatitis B virus carriers or individuals with chronic active hepatitis B or C, other chronic liver diseases, HIV infection,
6. Patients with abnormal liver function (ALT/AST 2 times higher); Moderate to severe renal impairment (glomerular filtration rate <60); hyperlipidemia not improved by lipid-lowering drugs,
7. Pregnant or lactating women,
8. Patients with a history of malignancy who do not meet the following condition (patients with malignant tumors who have been successfully treated for more than 5 years before screening without any evidence of recurrence),
9. Patients with previous visual field disorder or single eye dysfunction, cataract patients,
10. Patients with decompensated cardiac insufficiency or severe hypertension or diabetes mellitus, i.e. systolic blood pressure higher than 160mmhg or diastolic blood pressure higher than 100mmhg,
11. For patients with abnormal blood routine, lymphocytes <500/mm3 or ANC <1000/mm3 or HGB < 90g/L,
12. Patients with active bleeding and peptic ulcer,
13. Have used biological agents or added azathioprine, leflunomide, FK 506 within 1 month before enrollment,
14. Those who have participated in other drug clinical trials within 4 weeks,
15. Patients using CYP3A4 inhibitors or inducers such as ketoconazole, fluconazole, or rifampicin within 4 weeks.

Ages: 50 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with PMR-AS score <10 score at weeks 52 | at 52 weeks
  PMR-AS score: CRP (mg/dL)+Patient self-evaluation (0-10 visual scale)+ Physician global assessment (0-10 Visual Scale)+[morning stiffness (min) x0.1]+ EUL (0-3)

SECONDARY OUTCOMES:
PMR-AS score at weeks 24 | at 24 weeks
  PMR-AS score: CRP (mg/dL)+Patient self-evaluation (0-10 visual scale)+ Physician global assessment (0-10 Visual Scale)+[morning stiffness (min) x0.1]+ ability to elevate the upper limbs(EUL 0-3)
PMR-AS score at weeks 52 | at 52 weeks
  PMR-AS score: CRP (mg/dL)+Patient self-evaluation (0-10 visual scale)+ Physician global assessment (0-10 Visual Scale)+[morning stiffness (min) x0.1]+EUL (0-3)
CRP at weeks 24 | at 24 weeks
  CRP (mg/dL)
CRP at weeks 52 | at 52 weeks
  CRP (mg/dL)
ESR at weeks 24 | at 24 weeks
  ESR (mm/h)
ESR at weeks 52 | at 52 weeks
  ESR (mm/h)
Proportion of patients who discontinue drugs at weeks 52 | at 52 weeks
  Proportion of patients who discontinue Tof in the treatment group, prednisone in the control group at weeks 52

CONTACTS AND LOCATIONS:
Overall Officials: Weiqian Chen, Principal Investigator — Division of Rheumatology, the First Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Division of Rheumatology, the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Devauchelle-Pensec V, Carvajal-Alegria G, Dernis E, Richez C, Truchetet ME, Wendling D, Toussirot E, Perdriger A, Gottenberg JE, Felten R, Fautrel BJ, Chiche L, Hilliquin P, Le Henaff C, Dervieux B, Direz G, Chary-Valckenaere I, Cornec D, Guellec D, Marhadour T, Nowak E, Saraux A. Effect of Tocilizumab on Disease Activity in Patients With Active Polymyalgia Rheumatica Receiving Glucocorticoid Therapy: A Randomized Clinical Trial. JAMA. 2022 Sep 20;328(11):1053-1062. doi: 10.1001/jama.2022.15459. PMID 36125471
- [Background] Zhang L, Li J, Yin H, Chen D, Li Y, Gu L, Fu Y, Chen J, Chen Z, Yang S, Ye S, Li T, Lu L. Efficacy and safety of tofacitinib in patients with polymyalgia rheumatica: a phase 2 study. Ann Rheum Dis. 2023 May;82(5):722-724. doi: 10.1136/ard-2022-223562. Epub 2023 Jan 5. No abstract available. PMID 36604153
- [Background] Ma X, Yang F, Wu J, Xu B, Jiang M, Sun Y, Sun C, Yu Y, Xu D, Xiao L, Ren C, Chen C, Ye Z, Liang J, Lin J, Chen W. Efficacy and Safety of Tofacitinib in Patients with Polymyalgia Rheumatica (EAST PMR): An open-label randomized controlled trial. PLoS Med. 2023 Jun 29;20(6):e1004249. doi: 10.1371/journal.pmed.1004249. eCollection 2023 Jun. PMID 37384596
- [Background] Spinelli FR, Garufi C, Mancuso S, Ceccarelli F, Truglia S, Conti F. Tapering and discontinuation of glucocorticoids in patients with rheumatoid arthritis treated with tofacitinib. Sci Rep. 2023 Sep 20;13(1):15537. doi: 10.1038/s41598-023-42371-z. PMID 37730835
- [Background] Dejaco C, Kerschbaumer A, Aletaha D, Bond M, Hysa E, Camellino D, Ehlers L, Abril A, Appenzeller S, Cid MC, Dasgupta B, Duftner C, Grayson PC, Hellmich B, Hocevar A, Kermani TA, Matteson EL, Mollan SP, Neill L, Ponte C, Salvarani C, Sattui SE, Schmidt WA, Seo P, Smolen JS, Thiel J, Toro-Gutierrez CE, Whitlock M, Buttgereit F. Treat-to-target recommendations in giant cell arteritis and polymyalgia rheumatica. Ann Rheum Dis. 2024 Jan 2;83(1):48-57. doi: 10.1136/ard-2022-223429. PMID 36828585